CLINICAL TRIAL: NCT04885361
Title: A Randomized, Open Label, Phase 1 Study to Evaluate the Safety, Reactogenicity and Immunogenicity of OSE-13E, a Multiepitope-based Vaccine Candidate Against COVID-19, in Healthy Adults (COVEPIT-3)
Brief Title: To Evaluate the Safety, and Immunogenicity of Vaccine Candidate Against COVID-19, in Healthy Adults
Acronym: COVEPIT 3
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: OSE Immunotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSE-13E-C102
Record Dates: First submitted 2021-05-07; First posted 2021-05-13 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Coronavirus Disease (COVID-19)
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 injection (Experimental): The dose of 1 ml will be administered subcutaneously, preferably into deltoid region of the non-dominant arm.
  Interventions: Biological: CoVepiT (OSE13E)
- Arm 2 injections separated by 21 days (Experimental): The dose of 1 ml will be administered subcutaneously, preferably into deltoid region of the non-dominant arm.
  Interventions: Biological: CoVepiT (OSE13E)

INTERVENTIONS:
Biological: CoVepiT (OSE13E) — Study will be open label and will be randomized 1:1 in two parallel study arms receiving either one single dose or two doses separated by 21 days.

SUMMARY:
The proposed study is a phase 1 study which will evaluate the safety, reactogenicity and immunogenicity of two doses regimen of CoVepiT vaccine (OSE-13E) in the population of n=48 healthy volunteers 18 to 45 (inclusive) years old, vaccinated or not by authorized COVID-19 vaccine.

Study will be open label and will be randomized 1:1 in two parallel study arms receiving either one single dose or two doses separated by 21 days.

First 4 subjects will serve as sentinel cohort and 7 days reactogenicity data of these subjects will be reviewed by the independent safety monitoring committee (SMC) before proceeding to the vaccination of remaining volunteers. The progress of the study will be overviewed by a safety monitoring committee (SMC).

The CoVepiT vaccine is a peptide-based vaccine aiming to induce CD8+T-cell-mediated immune response against 11 different proteins of SARS-CoV-2 virus.

ELIGIBILITY:
Inclusion Criteria:

Subject's meeting all the following criteria are eligible to participate in this study:

* Males or females 18 to 45 (inclusive) years of age, at screening.
* Healthy participants as determined based on medical history, clinical laboratory results, vital sign measurements, and physical examination at screening.
* Subjects not previously vaccinated with any COVID-19 vaccine OR Subjects who have completed the vaccination according to an officially accepted scheme (e.g., healthcare workers), at least 4 weeks prior to enrollment, with an authorized vaccine which induces neutralizing antibodies against the SARS-CoV-2 Spike protein.
* Willing and able to give informed consent.
* Willing to accept following contraceptive measures:

Exclusion Criteria:

* Any ongoing, symptomatic acute or chronic illness requiring medical or surgical care, inclusive of changes in medication in the past 2 months (at the discretion of the investigator). This includes any current workup of undiagnosed illness that could lead to a new condition, including but not limited to any of the following conditions that are risk factors of severe illness from the virus that causes COVID-19:

  * Active cancer (malignancy) within 5 years prior to first study vaccination (with the exception of adequately treated non-melanomatous skin carcinoma, at the discretion of the investigator)
  * Chronic kidney disease
  * COPD
  * Moderate to severe asthma
  * Current tobacco smoking
  * People who have had an organ transplant.
  * Heart conditions, such as heart failure, coronary artery disease, or cardiomyopathies
  * BMI ≥ 30 kg/m2 or BMI <17 kg/m2
  * Type 2 diabetes mellitus
  * Chronic liver disease
  * Sickle cell disease Hypertension
* Type 1 diabetes
* Known infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBV).
* Participation in research involving an investigational product (drug/biologic/device) within 45 days prior to first study vaccination.
* History of a confirmed diagnosis of SARS, MERS or COVID-19 disease (confirmed by a specific test for each disease) or known exposure during 2-4 weeks prior to enrollment to a SARS-CoV-2 positive confirmed close contact (eg, family member, housemate, daycare provider, aged parent requiring care), at the discretion of the investigator.
* Professionals involved in direct care of the COVID-19 patients and with a high risk of exposure to SARS-CoV-2 (i.e., healthcare worker of intensive care unit at infectology department ).
* Currently taking any product (investigational or off-label) for prevention of COVID-19 disease.
* Positive rapid test for SARS-CoV-2 (ELISA or PCR) at screening or prior to first vaccination.
* Received influenza vaccination within 14 days prior to first study vaccination, or any other vaccine within 4 weeks prior to first study vaccination. NOTE: COVID-19 marketed vaccines may be allowed as long inclusion criterion #3 is met.
* Any autoimmune or immunodeficiency disease/condition (iatrogenic or congenital).
* Chronic administration (defined as more than 14 continuous days) of immunosuppressant, systemic glucocorticosteroids, or other immune-modifying drugs within 4 months prior to first study vaccination or anticipation of the need for immunosuppressive treatment within 6 months after last vaccination.
* Received immunoglobulin, blood-derived products, or other immunosuppressant drugs within 90 days prior to first study vaccination.
* Any acute illness concurrent or within 14 days prior to first study vaccination (medical history and/or physical examination) or documented temperature of ≥38°C during this period. This includes respiratory or constitutional symptoms consistent with SARS-CoV-2 (COVID-19) (ie, cough, sore throat, difficulty breathing)
* Known disturbance of coagulation (iatrogenic or congenital). NOTE: The use of ≤325 mg of aspirin per day as prophylaxis is permitted, but the use of other platelet aggregation inhibitors, thrombin inhibitors, Factor Xa inhibitors, or warfarin derivatives is exclusionary, regardless of bleeding history, because these imply treatment or prophylaxis of known cardiac or vascular disease.
* Any neurological disease or history of significant neurological disorder (eg, meningitis, seizures, multiple sclerosis, vasculitis, migraines, Guillain-Barré syndrome [genetic/congenital or acquired]).
* Vital sign (blood pressure, pulse, temperature) abnormalities of toxicity grade >1
* Clinical laboratory abnormalities of toxicity grade >1 for selected serum chemistry and hematology parameters
* Any known allergies to products contained in the investigational product or latex allergy, or history of severe allergic reaction (e.g., swelling of the mouth and throat, difficulty breathing, hypotension, or shock) that required medical intervention.
* Women who are pregnant, breastfeeding or who plan to become pregnant during the study.
* History of alcohol abuse or drug addiction within one year prior to the first study vaccination.
* Any condition that, in the opinion of the investigator, would pose a health risk to the subject if enrolled or could interfere with evaluation of the study vaccine or interpretation of study results (including neurologic or psychiatric conditions deemed likely to impair the quality of safety reporting).
* Study team member or first-degree relative of any study team member (inclusive of sponsor or delegate, and site personnel involved in the study).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-05-26 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of solicited local reactogenicity signs and symptoms | up to 7 days after each injection
The incidence of solicited systemic reactogenicity signs and symptoms | up to 7 days after each injection
The incidence of unsolicited adverse events in study participants. | up to 28 days after each vaccination.
The occurrence of serious adverse events (SAE). | throughout study completion, an average of 6 months.
The occurrence of adverse events of special interest (AESI), including potentially immune mediated disorders (pIMD) | throughout study completion, an average of 6 months.
Proportion of subjects with significantly increased CD8+ T cells responding to SARS-CoV-2 wild type epitopes at Week 6 - 1 versus 2 doses | Week 6

SECONDARY OUTCOMES:
Proportion of subjects with significantly increased CD8+ T cells responding to SARS-CoV-2 wild type epitopes | Day 22, Month 3 and Month 6
Geometric mean fold rise of CD8+ T cells responding to SARS-CoV-2 wild type | Day 22, Month 3 and Month 6
Proportion of participants achieving ≥2-fold rise of secreting spots specific to SARS-CoV-2 wild type epitopes | At baseline and after each vaccination
Change in geometric mean count (GMC) of CD8+ T cells antigen specific to SARS-CoV-2 wild type epitopes | from the pre-injection baseline (Day 1) to Day 22, Week 6, Month 3 and Month 6

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Vaccinology (CEVAC),, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided